CLINICAL TRIAL: NCT01614119
Title: Evaluation of the Cerebral Responses to Exercise in Hypoxia
Brief Title: Cerebral Responses During Exercise in Hypoxia
Acronym: CERVOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 1002; 2010-A00121-38 (Registry Identifier: ID RCB)
Record Dates: First submitted 2012-05-23; First posted 2012-06-07 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Brain Hypoxia; Hypoxia
Keywords: Cerebral; Oxygenation; Performance; Exercise
MeSH Terms: conditions — Hypoxia, Brain; Hypoxia; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sportsmen (Experimental): One single group of active healthy subjects was investigated
  Interventions: Other: Hypoxic exposure

INTERVENTIONS:
Other: Hypoxic exposure — Subjects breath either normoxic or hypoxic (FiO2 = 12%) gas mixture
  Other Names: Hypoxia (FiO2 = 12%)

SUMMARY:
While the exercise responses are classically described at the cardiorespiratory and muscle levels, recent data suggest that the brain is also significantly stressed by exercise and may even participate to performance limitation. In hypoxia in particular, cerebral responses to exercise may be altered and promote performance reduction during endurance exercise. In the present study, the investigators used innovative approaches to assess cerebral perturbations associated with exercise in hypoxia.

DETAILED DESCRIPTION:
In the classical paradigm of exercise physiology, cardio-respiratory capacity and muscle fatigue are though to set the limit of exercise tolerance. However, there are experimental situations where it is not possible to explain exercise performance limitation using this classical paradigm, and it is therefore necessary to look for an alternative. Recent investigations highlight changes associated with exercise in the brain, e.g. changes in cerebral perfusion, cerebral oxygenation and neuron excitability. Also, several results suggest that in some conditions, the central nervous system fails to drive the motoneurons adequately, i.e. the so called central fatigue. However, the phenomenon of central limitation to exercise and its underlying neurophysiological mechanisms are still to clarify. Cerebral metabolism and neurohumoral responses during fatiguing exercise are therefore to investigate in order to propose a new paradigm able to explain exercise limitation. Among the conditions where the classical paradigm of exercise performance limitation does not appear to suit the actual observations, exercise under hypoxic environment appears to be particularly challenging. Some data suggest indeed that the cerebral response to exercise may be substantially modified in hypoxia compared to normoxia.

Hence, in the present project, the investigators aim to evaluate the effect of hypoxia on brain adaptation to exercise in healthy human. In particular, the objective is to assess the brain neurophysiological response to a fatiguing exercise, including cerebral perfusion and oxygenation, cerebral activation, cortical excitability as well as the resultant motor command while inhaling normoxic or hypoxic gas mixtures. To fulfil these objectives, complementary methodological approaches will be used during exercise both normoxic and hypoxic conditions: functional magnetic resonance imaging (fMRI) will be used to evaluate cerebral activation, the perfusion imaging arterial spin labelling (ASL) nuclear magnetic resonance method will assess regional cerebral perfusion, near infrared spectroscopy (NIRS) will allow measurement of cerebral oxygenation, measurement of motor evoked potential in response to transcranial magnetic stimulation (TMS) will assess the cortical excitability, measurement of the level of central activation (assessed by TMS) and the electromyographic (EMG) signals will evaluate the motor command. Moreover, to account for the effect of the muscle mass involved during exercise and the duration of hypoxic exposure, brain adaptation to exercise in hypoxia will be assessed for motor task involving small (thumb adduction) or large (knee extension, cycle ergometry) muscle groups as well as for acute (<1 hour) or prolonged hypoxic exposure (several hours: 6 hours). This multi-technical approach will be possible through this collaborative project between three partners experts in brain function investigation and exercise physiology (Institut Fédératif de Recherche 'RMN Biomédical et Neurosciences' Joseph Fourier University and University Hospital, Grenoble; 'Exercise Physiology' Laboratory, University Hospital, St Etienne; 'Motor Efficiency and Deficiency Laboratory', Montpellier I University, Montpellier).

The investigators hypothesise that hypoxia would enhance the cerebral perturbation associated with a given fatiguing exercise, i.e. would induce greater reduction in cerebral blood and cerebral oxygenation, greater reduction in cortical excitability and central activation as well as larger reduction in central command, and this particularly when a large muscle mass is involved as well as when hypoxic exposure is prolonged.

This project aims to renew our vision of the limitation of human exercise performance as well as our understanding of exercise tolerance under hypoxemic conditions. The later is relevant for sport and altitude medicine dealing with exercise and altitude tolerance, as well as for diseases characterised by hypoxemia and exercise intolerance such as respiratory diseases like chronic obstructive pulmonary diseases for example.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-50 yrs
* No cardiovascular, respiratory or neuromuscular disorders

Exclusion Criteria:

* Cardiovascular, respiratory or neuromuscular diseases
* Contraindication for TMS and MRI

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in voluntary activation | Baseline and after 4h of exercise
  Maximum voluntary activation level measured using TMS

SECONDARY OUTCOMES:
Change in tissue oxygenation | Baseline and after 4 hours of exercise
  Muscle and cerebral oxygenation measured with NIRS and fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Wuyam, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France

REFERENCES:
- [Result] Verges S, Rupp T, Jubeau M, Wuyam B, Esteve F, Levy P, Perrey S, Millet GY. Cerebral perturbations during exercise in hypoxia. Am J Physiol Regul Integr Comp Physiol. 2012 Apr 15;302(8):R903-16. doi: 10.1152/ajpregu.00555.2011. Epub 2012 Feb 8. PMID 22319046